CLINICAL TRIAL: NCT00205530
Title: Evaluation of an Intervention Model for Family Crisis and Support (a Research Project Within the Traumatic Brain Injury Model System Grant)
Brief Title: Evaluation of an Intervention Model for Family Crisis and Support
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H133A02051604; H133A020516 (Other Grant/Funding Number: NIDRR); H133A070036 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Traumatic Brain Injury; Brain Injury, Chronic
Keywords: brain injury, family treatment
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injury, Chronic; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Brain Injury Family Intervention (BIFI) — The Brain Injury Family Intervention (BIFI) was developed over the last decade based upon considerable clinical experience and research review. The BIFI is a structured approach to helping families address their most common and salient issues, concerns, and challenges. The BIFI is implemented in five 90-minute sessions.
  Other Names: BIFI

SUMMARY:
To learn more about how a family treatment program helps people after brain injury. Specifically, do families feel better and function better after going through the program, and do patients feel better and function better after going through the program.

DETAILED DESCRIPTION:
To evaluate the efficacy of a structured outpatient family intervention program (BIFI) on family members' emotional well being, life satisfaction, needs, and family functioning; and to evaluate the impact of the BIFI on the emotional well being, life satisfaction, functional independence, vocational status, and neurobehavioral functioning of persons with acquired brain injury (ABI).

ELIGIBILITY:
Inclusion Criteria:

* Family members/caregiver friends and persons with acquired brain injury (ABI) who are at least three months postinjury. ABI is defined as damage to brain tissue caused by stroke, aneurysm, anoxia, or an external mechanical force as evidenced by: loss of consciousness, post traumatic amnesia (PTA), objective neurological findings, or skull fracture.

Exclusion Criteria:

* Families including individuals at imminent risk of psychiatric hospitalization, or in imminent danger of hurting themselves or others, as judged by the investigators.
* Individuals under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family members/caregiver friends and persons with ABI who are at least three months postinjury will be eligible to participate in the present investigation. ABI is defined as damage to brain tissue caused by stroke, aneurysm, anoxia, non-progressive brain tumor, infection, or an external mechanical force as evidenced by: loss of consciousness, post traumatic amnesia (PTA), objective neurological findings, or skull fracture. Penetrating wounds fitting the definition listed above will be included. Lacerations and/or bruises of the scalp or forehead without other criteria listed above will be excluded. All participants must be at least 18 years of age or older and able to understand and provide consent.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2003-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Family Needs Questionnaire (FNQ) | pre-treatment, post-treatment, 3 mo. follow-up
  The Family Needs Questionnaire (FNQ) is a widely used 40-item self-report questionnaire developed to measure family members' perceived needs after a family member sustains a brain injury. The items were designed to address diverse psychosocial and educational needs apparent in the acute and post-acute phases after injury. Family members rate the degree to which they perceive that each need has been met (not met, partly met, or met). A factor analytic investigation revealed six independent factors comprising six scales: Health Information, Emotional Support, Instrumental Support, Professional Support, Community Support Network, and Involvement with Care. The proportion of needs described as met (converted to a 10 point scale) was the primary family outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Kreutzer, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States